CLINICAL TRIAL: NCT00000925
Title: Evaluation of High Protein Supplementation in HIV-1-Positive Subjects With Stable Weight Loss
Brief Title: A Study to Evaluate High Protein Supplementation in HIV-Positive Patients With Stable Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 392; 11349 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; HIV Wasting Syndrome
Keywords: Dietary Proteins; HIV Wasting Syndrome
MeSH Terms: conditions — HIV Infections; HIV Wasting Syndrome

INTERVENTIONS:
Drug: Optimune oral nutritional supplement

SUMMARY:
The purpose of this study is to determine whether a high-quality protein food supplement will help HIV-positive patients maintain, and possibly gain, muscle mass.

Many HIV-positive patients lose weight that they are then unable to regain. This may be because patients are not eating enough protein or are not eating the right kinds of protein. The protein eaten in foods (such as meat, eggs, or beans) may not be able to make up for the amount of protein lost due to HIV infection. This study gives patients high-quality protein food supplements to help them maintain and/or gain weight.

DETAILED DESCRIPTION:
In many HIV-infected individuals with prior weight loss, the failure to regain weight and lean tissue is at least in part the consequence of inadequate protein intake or ingestion of a poor-quality protein rather than total caloric intake. Dietary sources of protein are presumably inadequate to meet the high metabolic needs caused by HIV infection. To achieve a target protein intake in the range (1.5 to 2.0 g/kg/day) demonstrated in other catabolic diseases necessary to achieve positive nitrogen balance and to generate substantial anabolic effects, this study will administer a supplement containing high-quality protein.

Two groups of 28 patients each are randomly chosen to receive either an oral nutritional supplement (Optimune) containing increased amounts of high-quality protein (whey), which is rich in cysteine and glutamine, or an isocaloric, identical-tasting supplement without added whey protein or amino acid supplementation. Weight, body composition, anthropometry, dietary intake, and general physical health are assessed at baseline and at Weeks 6 and 12. Plasma cysteine, glutathione, C-reactive protein, and prealbumin, along with urine IL-6, sTNFrII, and IL-1ra, are assessed at baseline and at Week 12.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are at least 18 years old.
* Have an HIV level less than 5,000 copies/ml within 30 days of study entry.
* Have lost weight in the past year, but your weight has remained fairly stable in the 2 months prior to enrollment.
* Are expected to live for at least 6 months.
* Are usually able to eat enough to maintain your present weight.
* Are able to complete a 3-day food diary.

Exclusion Criteria

You will not be eligible for this study if you:

* Have gained a significant amount of weight in the past 2 months.
* Have any opportunistic (HIV-associated) infections.
* Are unable to eat enough food for any reason, or are on tube feeding.
* Have nausea, diarrhea, or vomiting in the 14 days prior to study entry.
* Are being treated for diabetes.
* Are receiving chemotherapy or radiation therapy to treat cancer.
* Are pregnant or breast-feeding.
* Are allergic to milk or mangoes.
* Have an implanted defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 1999-05; Primary Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Mulligan, MD, Study Chair; Bruce R. Bistrian, MD, Study Chair; Fred R. Sattler, MD, Study Chair
Locations (19):
- United States (18):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of Cincinnati, Cincinnati, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Philadelphia Veterans Administration Med Ctr, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico